CLINICAL TRIAL: NCT05816044
Title: Evaluation of HALP Score in Preeclampsia
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, murat ibrahim toplu, medical doctor, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Other Study IDs: 67
Record Dates: First submitted 2023-04-01; First posted 2023-04-18 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Pre-Eclampsia
Keywords: preeclampsia; HALP score
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- preeclamptic pregnant woman
- healty preagnant woman

SUMMARY:
Preeclampsia is a serious condition that can occur during pregnancy and can pose problems for both the mother and the baby. It occurs in approximately 2-8% of all pregnancies globally and is caused by issues with blood vessels, leading to elevated blood pressure and other related health concerns. Additionally, insufficient nutrition and inflammation within the mother's body may contribute to the development of preeclampsia.

The HALP score serves as a tool to assess various elements within the blood, indicating inflammation or inadequate nutrition. Although it has been utilized in other medical contexts, its application during pregnancy remains limited. The HALP score has been employed to predict the emergence of ailments such as heart disease and cancer. Given that preeclampsia can stem from inflammation and poor nutrition, the potential of the HALP score in predicting the likelihood of preeclampsia during pregnancy is being examined through research.

DETAILED DESCRIPTION:
Preeclampsia is a hypertensive disorder affecting multiple body systems that poses a risk of maternal and fetal morbidity and mortality. The global prevalence of preeclampsia is estimated to be around 2-8% of all pregnancies. The pathophysiology of preeclampsia is complex and involves endothelial dysfunction and vasospasm, resulting in hypertension and end-organ damage. The development of preeclampsia is influenced by various factors, including abnormalities in the placenta, genetic factors, and maternal immune system. In addition, poor maternal nutrition and inflammation have also been identified as potential contributors to the development of preeclampsia.

The HALP score is a composite measure of hemoglobin, albumin, lymphocyte, and platelet parameters that has been suggested as a possible indicator of systemic inflammation and malnutrition. Although the HALP score has not been extensively studied in obstetrics, it has been investigated in various medical fields as a predictor of adverse outcomes such as cardiovascular disease and cancer. Given the significance of inflammation and malnutrition in the development of preeclampsia, it is important to investigate the potential usefulness of the HALP score in predicting this condition.

Due to the limited research on the application of the HALP score in obstetrics and the possible role of inflammation and malnutrition in the pathogenesis of preeclampsia, a retrospective study is being planned to explore the potential utility of the HALP score as a predictor of preeclampsia. By analyzing the relationship between the HALP score and the development of preeclampsia, valuable insights can be obtained regarding the potential involvement of inflammation and malnutrition in the development of this disorder.

ELIGIBILITY:
Inclusion Criteria:

* in preeclampsia group

  * Having a singleton pregnancy.
  * Pregnant women diagnosed with preeclampsia according to the American College of Obstetricians and Gynecologists (ACOG) 2020 gestational hypertension and preeclampsia bulletin criteria.
  * Pregnant women who do not have a systemic inflammatory disease other than preeclampsia
  * Pregnant women whose delivery and postpartum follow-up are in our clinic
* In the Control Group

  * Having a singleton pregnancy
  * Pregnant women who have no history or signs of systemic disease
  * Pregnant women who have not found any maternal or fetal abnormality in the pregnancy follow-up
  * Pregnant women whose delivery and postpartum follow-up are in our clinic

Exclusion Criteria:

* Multiple gestation pregnancies
* Known chronic or systemic disease (hypo or hyperthyroidism, diabetes, chronic hypertension, heart diseases, hyperlipidemia, chronic liver failure, acute or chronic kidney failure, etc.)
* Unknown pregnancy follow-up or fetal or maternal abnormalities detected during follow-up pregnant women
* Pregnant women whose delivery or postpartum follow-up is outside of our clinic

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study is a case-control retrospective study. Pregnant women between the ages of 18-44 who were diagnosed with preeclampsia and healthy pregnant woman in our clinic and whose follow-up and birth were in our hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
evaluate the HALP score in preeclamptic and healty pregnant woman | From January 2021 to January 2023, examination findings and medical tests of pregnant women diagnosed with preeclampsia, as well as healthy pregnant women, will be retrospectively evaluated by utilizing data documented by scanning patient records.
  The HALP score, which comprises Hemoglobin, Albumin, Lymphocyte, and Platelet parameters, is a useful tool for healthcare professionals to evaluate the nutritional and inflammatory status of a patient. Higher HALP scores are indicative of better immune-nutritional function, whereas lower scores suggest poorer immune-nutritional status. Thus, the HALP score provides valuable prognostic information that can guide treatment decisions and risk stratification for patients with various medical conditions. Currently, there is no standardized or universally accepted cutoff for the HALP score to predict specific outcomes. The optimal threshold for the HALP score is disease-specific and largely dependent on the study. This is based on the available literature.

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Dr. Cemil Taşcıoğlu City Hospital, Istanbul, Turkey (Türkiye)